CLINICAL TRIAL: NCT02010736
Title: Immediate Effects of a Single Treadmill Gait Training Session With Additional Loading on Kinematic Gait Parameters in Children With Spastic Cerebral Palsy
Brief Title: Loading Gait in Spatic Cerebral Palsy
Acronym: SCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Ana Raquel Rodrigues Lindquist, PhD, Universidade Federal do Rio Grande do Norte
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP-UFRN 76519/2012
Record Dates: First submitted 2013-12-05; First posted 2013-12-13 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Spastic Hemiplegic Cerebral Palsy
Keywords: Cerebral palsy; Gait; Weight Bearing; Rehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spastic Hemiparetic Cerebral Palsy (Experimental): Single treadmill gait training with additional loading
  Interventions: Other: Single treadmill gait training with additional loading

INTERVENTIONS:
Other: Single treadmill gait training with additional loading

SUMMARY:
The purpose of this study is to observe the behavior of kinematic variables in children with spastic hemiparetic cerebral palsy (SHCP), immediately after treadmill gait training with ankle loading.

The children underwent a single treadmill training session with ankle loading. The kinematic parameters were assessed in three phases: before training (PRE); immediately after training (POST); and 5 minutes after the end of training (FOLLOW UP).

The investigators hypothesized that the treadmill gait training with additional lower limb loading would be a disturbance capable of modifying the locomotor strategy of children with SHCP, by the increase in kinematic parameters in the swing phase of gait.

ELIGIBILITY:
Inclusion Criteria:

* Spastic Hemiparetic Cerebral Palsy;
* Being able to walk without an assistive device (levels I or II of the Gross Motor Function Classification System - GMFCS);
* Not having undergone muscle lengthening surgery within the previous year;
* Not having applied botulin toxin to the lower limbs or serial casting in the previous 6 months.

Exclusion Criteria:

* Inability to understand simple commands to perform the training and evaluation;
* Inability to walk on the treadmill with or without load on the lower limbs;
* Presence of any physical pain or discomfort during the course of training.

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Changes in kinematic gait parameters after treadmill trainning with ankles loading | Immediately after training with ankles loading (POST phase)
  Kinematic gait data were captured by Qualisys Track Manager 1.6.0.x - QTM software and exported to Visual3D processing software, to reconstruct the segments and create a biomechanical model. It was carried out in two stages: static and dynamic collection. The dynamic collection was performed while the children walked on the electric treadmill.
  The primary outcome measure was the following spatiotemporal variables at the POST phase: cadence (steps/min), stride length (m), paretic step length (m), stance time (%), swing time (%) paretic lower limb (PLL), double stance (%), symmetry ratio and stance/swing time ratio. With respect to angular variables, the following parameters was analysed: angular displacement (maximum flexion, maximum extension and range of motion) of the hip and knee were investigated (º).

SECONDARY OUTCOMES:
Changes in kinematic gait parameters after five minutes of rest | After five minutes of rest (FOLLOW UP phase)
  Kinematic gait data were captured by Qualisys Track Manager 1.6.0.x - QTM software and exported to Visual3D processing software, to reconstruct the segments and create a biomechanical model. It was carried out in two stages: static and dynamic collection. The dynamic collection was performed while the children walked on the electric treadmill.
  The secundary outcome measure was the same spatiotemporal and angular variables investigated at the POST phase although in this condition they was analysed at FOLLOW UP phase.

CONTACTS AND LOCATIONS:
Overall Officials: Camila R Simão, MSc, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (1):
- Universidade Federal do Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil

REFERENCES:
- See also: Cerebral palsy — http://vsearch.nlm.nih.gov/vivisimo/cgi-bin/query-meta?v%3Aproject=medlineplus&query=cerebral+palsy&x=10&y=9
- See also: Gait training — http://vsearch.nlm.nih.gov/vivisimo/cgi-bin/query-meta?v%3Aproject=medlineplus&query=gait+training&x=14&y=21